CLINICAL TRIAL: NCT04706156
Title: Oral Side Effects of COVID-19 Vaccine: A Multicenter Cross-sectional Study
Brief Title: Oral Side Effects of COVID-19 Vaccine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Masaryk University (Other)
Collaborators: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other); University of Giessen (Other); University of Kiel (Other); Yeditepe University (Other)
Responsible Party: Sponsor
Other Study IDs: OSECV
Record Dates: First submitted 2021-01-11; First posted 2021-01-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-01

CONDITIONS: Oral Manifestations; Covid19; Vaccine Adverse Reaction
Keywords: COVID19; Oral Manifestations; Vaccine Adverse Reaction
MeSH Terms: conditions — Oral Manifestations; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Vaccinated Healthcare Workers (CZ): Czech healthcare workers who received COVID-19 vaccine during the last 30 days (n=385)
  Interventions: Biological: COVID-19 Vaccine
- Vaccinated Healthcare Workers (DE): German healthcare workers who received COVID-19 vaccine during the last 30 days (n=385)
  Interventions: Biological: COVID-19 Vaccine
- Vaccinated Healthcare Workers (SK): Slovak healthcare workers who received COVID-19 vaccine during the last 30 days (n=385)
  Interventions: Biological: COVID-19 Vaccine
- Vaccinated Healthcare Workers (TR): Turkish healthcare workers who received COVID-19 vaccine during the last 30 days (n=385)
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — Receiving coronavirus disease (COVID-19) vaccine e.g. Pfizer-BioNTech, Moderna, Oxford/AstraZeneca, or Sinovac COVID-19 Vaccine

SUMMARY:
This study is a multicenter cross-sectional survey-based study conducted in four European countries (Czech Republic, Germany, Slovak Republic, and Turkey). An online questionnaire will be utilized to collect data from volunteer subjects following the STROBE reporting guidelines of cross-sectional studies.

DETAILED DESCRIPTION:
The primary objective of this multicentre cross-sectional survey-based study is to estimate the prevalence of oral side effects of COVID-19 vaccine in the short term.

The secondary objectives are:

* to identify the risk factors of COVID-19 vaccine oral side effects in the short term.
* to evaluate the relationship between oral side effects and other inflammatory side effects of COVID-19 vaccine in the short term.

The target population is healthcare workers as they are identified among the priority groups of COVID-19 vaccine deployment plans in the EU/EEA and the UK. One more reason to select the healthcare workers among different groups of the population, their higher awareness about the possible vaccine-related oral side-effects so that more accurate and reliable results can be obtained.

A self-administered questionnaire will be developed, and its content validity will be tested using a panel of experts. The test re-test reliability of the questionnaire will be tested by 30 volunteers (10 Czech, 10 Turkish, 10 German) to achieve at least a Cronbach's alpha of 0.70. The questionnaire will be available in five languages; Czech, English, German, Slovak and Turkish. Dual forward translation and expert panels will produce equivalent Czech, German, Slovak and Turkish versions of the questionnaire.

The questionnaire will be composed of multiple-choice items divided into four main categories; a) demographic data including gender, age, location of practice, profession, and experience, b) medical anamnesis including medical comorbidities, medications, and recent oral symptoms, c) COVID-19 related anamnesis including vaccination date, previous infection, and exposure to infected cases, and d) vaccine side effects including inflammatory symptoms, cutaneous symptoms, and oral symptoms. (Annex 1)

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers who received COVID-19 vaccine during the last 30 days.
* Participating subjects should be at least 18-year-old and able to give their informed consent independently.

Exclusion Criteria:

* The healthcare workers who did not receive the COVID-19 vaccine recently.
* Non-healthcare workers who received the COVID-19 vaccine recently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population is healthcare workers as they are identified among the priority groups of COVID-19 vaccine deployment plans in the EU/EEA and the UK. One more reason to select the healthcare workers among different groups of the population, their higher awareness about the possible vaccine-related oral side-effects so that more accurate and reliable results can be obtained.
Sampling Method: Non-Probability Sample
Enrollment: 1540 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Oral Side Effects | 0-30 days after the COVID-19 vaccine shot
  Dichotomous outcome for the emergence of oral side effects (e.g. ulcers, vesicles, blisters, plaque, mouth odour, bleeding gum, burning gingiva, etc) following receiving the COVID-19 vaccine.

SECONDARY OUTCOMES:
Dermatologic Side Effects | 0-30 days after the COVID-19 vaccine shot
  Dichotomous outcome for the emergence of dermatologic side effects (e.g. injection site swelling, or redness, rash, urticaria, angioedema, etc) following receiving the COVID-19 vaccine.
General (common) Side Effects | 0-30 days after the COVID-19 vaccine shot
  Dichotomous outcome for the emergence of typical side effects (e.g. injection site pain, injection site swelling, injection site redness, tiredness, headache, nausea, muscle pain, joint pain, fever, swollen lymph nodes (lymphadenopathy), etc) following receiving the COVID-19 vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Abanoub Riad, DDS, Principal Investigator — Masaryk University
Locations (4):
- Department of Public Health, Faculty of Medicine, Masaryk University, Brno, South-Moravia, Czechia
- Germany (2):
  - Department of Cranio-Maxillofacial Surgery, Justus-Liebig University Giessen, Giessen, Hesse
  - Clinic for Conservative Dentistry and Periodontology, School of Dental Medicine, Christian-Albrecht's University, Kiel, Schleswig-Holstein
- Department of Maxillofacial Surgery, F. D. Roosevelt University Hospital, Banská Bystrica, Banská Bystrica Region, Slovakia

IPD SHARING:
Plan to Share IPD: No
In accordance with the General Data Protection Regulation (GDPR), the data controller is Masaryk University (MUNI) and will be used solely by MUNI for the purpose of research in area of public health. The collected data will not be accessed or used by other institutions or for any other purposes. The data will be processed and analysed during the duration of the project (approximately one year). After the project is finished, the data will be encrypted and safely stored by MU as a measure to secure the integrity of the research.

REFERENCES:
- [Background] Riad A, Klugar M, Krsek M. COVID-19-Related Oral Manifestations: Early Disease Features? Oral Dis. 2022 Apr;28 Suppl 1(Suppl 1):940-942. doi: 10.1111/odi.13516. Epub 2020 Jul 16. No abstract available. PMID 32603497
- [Background] Riad A, Gad A, Hockova B, Klugar M. Oral candidiasis in non-severe COVID-19 patients: call for antibiotic stewardship. Oral Surg. 2022 Aug;15(3):465-466. doi: 10.1111/ors.12561. Epub 2020 Oct 9. No abstract available. PMID 33042219
- [Background] Riad A, Kassem I, Stanek J, Badrah M, Klugarova J, Klugar M. Aphthous stomatitis in COVID-19 patients: Case-series and literature review. Dermatol Ther. 2021 Jan;34(1):e14735. doi: 10.1111/dth.14735. Epub 2021 Jan 10. No abstract available. PMID 33389769
- [Background] Riad A, Kassem I, Hockova B, Badrah M, Klugar M. Halitosis in COVID-19 patients. Spec Care Dentist. 2021 Mar;41(2):282-285. doi: 10.1111/scd.12547. Epub 2020 Nov 29. No abstract available. PMID 33249615
- [Background] Riad A, Kassem I, Badrah M, Klugar M. The manifestation of oral mucositis in COVID-19 patients: A case-series. Dermatol Ther. 2020 Nov;33(6):e14479. doi: 10.1111/dth.14479. Epub 2020 Nov 8. No abstract available. PMID 33125803
- [Background] Riad A, Kassem I, Issa J, Badrah M, Klugar M. Angular cheilitis of COVID-19 patients: A case-series and literature review. Oral Dis. 2022 Apr;28 Suppl 1(Suppl 1):999-1000. doi: 10.1111/odi.13675. Epub 2020 Oct 23. No abstract available. PMID 33043573
- [Background] Riad A, Kassem I, Hockova B, Badrah M, Klugar M. Tongue ulcers associated with SARS-CoV-2 infection: A case series. Oral Dis. 2022 Apr;28 Suppl 1:988-990. doi: 10.1111/odi.13635. Epub 2020 Sep 25. No abstract available. PMID 32889763
- [Background] Riad A, Kassem I, Badrah M, Klugar M. Acute parotitis as a presentation of COVID-19? Oral Dis. 2022 Apr;28 Suppl 1:968-969. doi: 10.1111/odi.13571. Epub 2020 Aug 6. No abstract available. PMID 32713097
- [Background] Riad A, Kassem I, Badrah M, Klugar M. COVID-19 transient snoring (CVTS): Clinical and laboratory description. J Med Virol. 2021 Apr;93(4):1890-1892. doi: 10.1002/jmv.26705. Epub 2020 Dec 17. No abstract available. PMID 33289127
- See also: Effects of the Influenza Vaccine on the Oral Cavity — https://stars.library.ucf.edu/cgi/viewcontent.cgi?article=1306&context=honorstheses
- See also: Annex 1 — https://muni.cz/go/osecv